CLINICAL TRIAL: NCT03948802
Title: Evaluation of Interleukin 33 in Relation to Selected Inflammatory Parameters in Patients With the Acute Ischemic Stroke of the Brain
Brief Title: Evaluation of IL-33 in Patients With the Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Jan Biziel University Hospital No 2 in Bydgoszcz (Other)
Responsible Party: Principal Investigator, Pawel Sokal, Head of Department of Neurosurgery and Neurology, Jan Biziel University Hospital No 2 in Bydgoszcz
Other Study IDs: JBUH-NN-STROKE-IL33
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; Interleukin 33; ASTRAL; DRAGON; NIHSS
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For the examination a venous blood is taken up from the elbow vein - 10 ml into the test tube containing 3.2 % solution of sodium citrate, for routine examinations (including the morphology with the smear, hsCRP). The concentration of interleukin 33 is assessed with the Elisa test. Blood is taken twice: in first twenty-four hours and seventh day after the cerebral stroke.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STROKE GROUP: Cerebral ischemic stroke patients treated.
  Interventions: Diagnostic Test: Interleukine 33 test in blood plasma
- CONTROL GROUP: Ambulatory healthy patients
  Interventions: Diagnostic Test: Interleukine 33 test in blood plasma

INTERVENTIONS:
Diagnostic Test: Interleukine 33 test in blood plasma — ELISA test for Interleukin 33

SUMMARY:
Aim of the study is to evaluate the usefulness of interleukin 33 in the blood plasma in patients with the acute ischemic stroke of the brain in relation to mode of treatment (thrombolysis, thrombectomy, no treatment), risk factors in correlation with other inflammatory state markers (hsCRP, morphology with smear ). Blood is collected on the first and seventh days of stroke.

The purpose is to clarify utility of IL 33 as a biomarker of acute stroke.

DETAILED DESCRIPTION:
Stroke is the third most frequent cause of death in highly developed countries (after heart disease and cancer), the main cause of disability in adults and the second most frequent cause of dementia syndromes. The annual incidence of stroke in the general population is approximately 0.2%. The risk of stroke increases with age.

Globally 15 million people are affected each year and 5.5 million die every year for this reason (20% in 30 days and up to 40% in a year from getting ill). In Poland, the incidence of stroke is around 175/100,000 in men and 125/100 in women.It is assumed that the cause of sudden cerebral insufficiency is mainly the embolism coming from the newly formed wall clot forming at the site of the atherosclerotic plaque rupture.

In recent years, the role of inflammatory factors is associated with the occurrence of severe atherosclerotic complications such as stroke or heart attack. Cytokines are glycoproteins that are released by activated cells of various tissues. They have a significant impact on the inflammation processes, they control all phases of the immune response. Interleukin is one of the cytokine groups. This study aims to find a relationship between level of IL 33 concentration and the size of the stroke and neurological deficit.

Blood will be collected on the first and seventh days of stroke for examination of Il 33, blood morphology and hsCRP

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Consent on participation
* Diagnosed Ischemic Stroke

Exclusion Criteria:

* Active cancer disease
* Kidney failure
* Liver failure
* Pregnancy
* Breastfeeding

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with ischemic stroke
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
NIHSS The National Institutes of Health Stroke Scale | 7 days
  Score 0-6 gently course of the cerebral stroke more than 6 increased manifestations of the cerebral infarction.Patients will be assessed before and after the trial to compare how each participant improved after given the intervention.
DRAGON scale | 7 days
  Comparison of patients in DRAGON scale on the 1st and the 7th day. DRAGON scale was developed to make early predictions about clinical outcomes for ischemic stroke patients using only information that is available shortly after they arrive at the hospital and before tPA is given. The DRAGON score, especially at the low and high end of the scale, can help predict which patients are likely to have good clinical outcomes and those who are likely to have miserable clinical outcomes even if given tPA. These patients may also be potential candidates for endovascular thrombectomy, though the benefits of this procedure have not yet been demonstrated in the literature.
ASTRAL scale | 1 day
  ASTRAL scale is used in patients with acute ischemic stroke admitted within 24 hours of stroke onset. It can provide additional information on medium-term functional outcome in patients that have suffered acute ischemic stroke, in addition to clinical judgment based on relevant clinical and laboratory variables.It can be used to adjust for functional outcome in multivariate models in acute stroke-related research studies.It can serve as a selection criterion for cohorts in acute stroke-related research studies.
Modified Rankin Scale | 7 days
  Change in disability. mRS can help users determine the degree of disability in patients who have suffered a stroke. mRS assesses disability in patients who have suffered a stroke and is compared over time to check for recovery and degree of continued disability. A score of 0 is no disability, 5 is disability requiring constant care for all needs; 6 is death
IL 33 and hsCRP concentration | 7 days
  Evaluation of IL 33 and hsCRP concentration, morphology with smear on the first and seventh day.

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Sokal, Principal Investigator — Jan Biziel University Hospital Collegium Medicum Nicolaus Copernicus University
Locations (1):
- Jan Biziel University Hospital nr 2 Collegium Medicum Nicolaus Copernicus University, Bydgoszcz, Poland

IPD SHARING:
Plan to Share IPD: No